CLINICAL TRIAL: NCT06412991
Title: Implementing Cycling as a Mobility Option for Operative and Non-operative Patients With Small Bowel Obstruction and Ileus Admitted by Northeast Acute Care Surgery at Atrium Health Cabarrus
Brief Title: Pedal Movement - Implementing Cycling as a Mobility Option
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00111263
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-05

CONDITIONS: Ileus
Keywords: bowel function; bowel obstruction; cycle therapy; mobility
MeSH Terms: conditions — Ileus; Intestinal Obstruction

STUDY DESIGN:
Intervention Model Description: Any patient admitted to the NorthEast Acute Care Surgery service on the Post Surgical Care 1 unit diagnosed with ileus, non-operative small bowel obstruction, or has had bowel surgery and with post operative small bowel obstruction and/or ileus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycle therapy (Experimental): The patient will either ambulate a short distance to recumbent bike which will be stored on the postsurgical 1 unit or be assisted out of bed to use floor cycle bike. After the patient demonstrates individual competency with either cycle modality, the patient may participate in this activity with nursing staff but will not require Physical Therapy (PT) presence at the time of use. This will allow the patient to participate multiple times a day if they choose.
  Interventions: Behavioral: Cycle Therapy
- ambulation as mobilization modality (No Intervention): ambulation by surgical team

INTERVENTIONS:
Behavioral: Cycle Therapy — The patient will either ambulate a short distance to recumbent bike which will be stored on the postsurgical 1 unit or be assisted out of bed to use floor cycle bike.
  Arms: Cycle therapy

SUMMARY:
Cycling has been a proven exercise for decades as a low impact option to strengthen the lower body and improve cardiovascular health. There is also evidence that cycling helps to stimulate the contraction of the muscles in the intestine. Other outcomes frequently examined when considering benefits of ambulation include decreased rates of venous thromboembolic events, pneumonia, and decreased hospital length of stays. Therefore, there is added value to consider alternate mobility modalities.

DETAILED DESCRIPTION:
Ileus is a common post operative occurrence, one that not only causes patient discomfort but also contributes to considerable economic impact and can potentially progress to other serious complications. Historically ileus has been difficult to define. Review of the literature produces a general definition to include a varying time frame upon which a patient is not tolerating an oral diet, unable to pass flatus or stool, symptoms of nausea, vomiting, and sometimes abdominal pain. Small bowel obstruction, while different pathophysiology than ileus, presents similar manifestations. Often ileus and small bowel obstruction follow the same pathway aimed at attempted resolution with attempts at conservative management. Efforts to resolve ileus and nonoperative small bowel obstruction include bowel rest, nasogastric decompression, and encouraging mobility. Many studies support the practice of mobilization through ambulation as an effort to encourage return of bowel function. What is lacking in review of the literature however are other modalities to offer the patient in efforts to assist and encourage patients to mobilize outside of ambulation.

ELIGIBILITY:
Inclusion Criteria:

* Admission to NorthEast Acute Care Surgery
* Admitted on Post Surgical Care 1 unit
* Diagnosis of small bowel obstruction
* Diagnosis of ileus
* Any patient that has had intestinal surgery
* Age 18-90

Exclusion Criteria:

* Age < 18
* Pregnancy
* Incarceration
* Non-English speaking

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Length of time to first Bowel Movement (BM) | Day 30
  Length of time to first Bowel Movement
Length of time to first flatus | Day 30
  Length of time to first flatus

SECONDARY OUTCOMES:
Rates of Venous thromboembolism (VTE) | Day 30
  VTE occurrence within 30 days post discharge
Rates of pneumonia | Day 30
  Pneumonia occurrence within 30 days post discharge
Hospital length of stay | Day 30
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Mallory Royall, NP, DNP, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Northeast Acute Care Surgery, Concord, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT06412991/ICF_000.pdf